CLINICAL TRIAL: NCT07293897
Title: A Cohort Study to Investigate the Risk of Liver Disorder of Livmarli Oral Solution in Patients With Japan Alagille Syndrome (ALGS) and Progressive Familial Intrahepatic Cholestasis (PFIC) Registered in the Comprehensive and Informative Registry System for Childhood Liver Disease (CIRCLe)
Brief Title: A Database Study of Maralixibat (TAK-625) in Participants With Alagille Syndrome (ALGS) and Progressive Familial Intrahepatic Cholestasis (PFIC)
Status: Not yet recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-625-4002
Record Dates: First submitted 2025-12-17; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Alagille Syndrome (ALGS); Progressive Familial Intrahepatic Cholestasis (PFIC)
Keywords: Alagille Syndrome (ALGS); Progressive Familial Intrahepatic Cholestasis (PFIC)
MeSH Terms: conditions — Alagille Syndrome; Cholestasis, progressive familial intrahepatic 1 | interventions — maralixibat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Alagille Syndrome (ALGS) Group: Participants with Alagille Syndrome (ALGS) who received maralixibat in accordance with package insert.
  Interventions: Drug: Maralixibat
- Progressive Familial Intrahepatic Cholestasis (PFIC) Group: Participants with Progressive Familial Intrahepatic Cholestasis (PFIC) who received maralixibat in accordance with package insert.
  Interventions: Drug: Maralixibat

INTERVENTIONS:
Drug: Maralixibat — Maralixibat Oral Solution 10 milligrams (mg)/milliliters (mL)
  Other Names: TAK-625; Livmarli Oral Solution

SUMMARY:
This study is a database study in Japan for maralixibat (TAK-625) used to treat participants with Alagille Syndrome (ALGS) and Progressive Familial Intrahepatic Cholestasis (PFIC).

The main aim of the study is to evaluate the risk of liver disorder during the use of maralixibat in Japanese patients with ALGS or PFIC.

This database study will conduct in use of medical database called Comprehensive and Informative Registry system for Childhood Liver Disease (CIRCLe).

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of ALGS or PFIC within the enrollment period.
* There is a prescription for Livmarli during the enrollment period (Index date: the date of the first prescription within the enrollment period).

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of this study are all participants who meet the inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01-09 (Estimated); Primary Completion 2031-06-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with ALGS who Experience Liver Disorder Evaluated with Outcome Definition 1 (Side Effects) | Up to 6 years as data period
  Percentage of participants with ALGS who will experience liver disorder will be reported. Outcome Definition 1 (side effects) will be used to estimate this outcome measure. Outcome Definition 1 (side effects) will define as follows: For the adverse event entry form, if all of the following conditions are met, it is defined as "liver disorder". (1) "Maralixibat (Livmarli)" has been selected as the drug to be administered. (2) "Yes" is selected for the presence or absence of adverse events due to the administered drug. (3) "Liver impairment and liver failure" are selected as symptoms/findings due to the administered drugs. (4) Date of occurrence or discovery of adverse event within the follow-up period. (5) "Unlikely" or "Not related" was not selected for the association between this adverse event and the treatment.
Percentage of Participants with PFIC who Experience Liver Disorder Evaluated with Outcome Definition 1 (Side Effects) | Up to 6 years as data period
  Percentage of participants with PFIC who will experience liver disorder will be reported. Outcome Definition 1 (side effects) will be used to estimate this outcome measure. Outcome Definition 1 (side effects) will define as follows: For the adverse event entry form, if all of the following conditions are met, it is defined as "liver disorder". (1) "Maralixibat (Livmarli)" has been selected as the drug to be administered. (2) "Yes" is selected for the presence or absence of adverse events due to the administered drug. (3) "Liver impairment and liver failure" are selected as symptoms/findings due to the administered drugs. (4) Date of occurrence or discovery of adverse event within the follow-up period. (5) "Unlikely" or "Not related" was not selected for the association between this adverse event and the treatment.
Time to Onset of Liver Disorder in Participants with ALGS Evaluated with Outcome Definition 1 (Side Effects) | Up to 6 years as data period
  Time to onset of liver disorder in participants with ALGS will be reported. Outcome Definition 1 (side effects) will be used to estimate this outcome measure. Outcome Definition 1 (side effects) will define as follows: For the adverse event entry form, if all of the following conditions are met, it is defined as "liver disorder". (1) "Maralixibat (Livmarli)" has been selected as the drug to be administered. (2) "Yes" is selected for the presence or absence of adverse events due to the administered drug. (3) "Liver impairment and liver failure" are selected as symptoms/findings due to the administered drugs. (4) Date of occurrence or discovery of adverse event within the follow-up period. (5) "Unlikely" or "Not related" was not selected for the association between this adverse event and the treatment.
Time to Onset of Liver Disorder in Participants with PFIC Evaluated with Outcome Definition 1 (Side Effects) | Up to 6 years as data period
  Time to onset of liver disorder in participants with PFIC will be reported. Outcome Definition 1 (side effects) will be used to estimate this outcome measure. Outcome Definition 1 (side effects) will define as follows: For the adverse event entry form, if all of the following conditions are met, it is defined as "liver disorder". (1) "Maralixibat (Livmarli)" has been selected as the drug to be administered. (2) "Yes" is selected for the presence or absence of adverse events due to the administered drug. (3) "Liver impairment and liver failure" are selected as symptoms/findings due to the administered drugs. (4) Date of occurrence or discovery of adverse event within the follow-up period. (5) "Unlikely" or "Not related" was not selected for the association between this adverse event and the treatment.

SECONDARY OUTCOMES:
Percentage of Participants with ALGS who Experience Liver Disorder Evaluated with Outcome Definition 2 (Adverse Events) | Up to 6 years as data period
  Percentage of participants with ALGS who will experience liver disorder will be reported. Outcome Definition 2 (Adverse Events) will be used to estimate this outcome measure. Outcome Definition 2 (Adverse Events) will define as follows: For the adverse event entry form, if all of the following conditions are met, it is defined as "liver disorder". (1) "Maralixibat (Livmarli)" has been selected as the drug to be administered. (2) "Yes" is selected for the presence or absence of adverse events due to the administered drug. (3) "Liver impairment and liver failure" are selected as symptoms/findings due to the administered drugs. (4) Date of occurrence or discovery of adverse event within the follow-up period.
Percentage of Participants with PFIC who Experience Liver Disorder Evaluated with Outcome Definition 2 (Adverse Events) | Up to 6 years as data period
  Percentage of participants with PFIC who will experience liver disorder will be reported. Outcome Definition 2 (Adverse Events) will be used to estimate this outcome measure. Outcome Definition 2 (Adverse Events) will define as follows: For the adverse event entry form, if all of the following conditions are met, it is defined as "liver disorder". (1) "Maralixibat (Livmarli)" has been selected as the drug to be administered. (2) "Yes" is selected for the presence or absence of adverse events due to the administered drug. (3) "Liver impairment and liver failure" are selected as symptoms/findings due to the administered drugs. (4) Date of occurrence or discovery of adverse event within the follow-up period.
Time to Onset of Liver Disorder in Participants with ALGS Evaluated with Outcome Definition 2 (Adverse Events) | Up to 6 years as data period
  Time to onset of liver disorder in participants with ALGS will be reported. Outcome Definition 2 (adverse events) will be used to estimate this outcome measure. Outcome Definition 2 (adverse events) will define as follows: For the adverse event entry form, if all of the following conditions are met, it is defined as "liver disorder". (1) "Maralixibat (Livmarli)" has been selected as the drug to be administered. (2) "Yes" is selected for the presence or absence of adverse events due to the administered drug. (3) "Liver impairment and liver failure" are selected as symptoms/findings due to the administered drugs. (4) Date of occurrence or discovery of adverse event within the follow-up period.
Time to Onset of Liver Disorder in Participants with PFIC Evaluated with Outcome Definition 2 (Adverse Events) | Up to 6 years as data period
  Time to onset of liver disorder in participants with PFIC will be reported. Outcome Definition 2 (adverse events) will be used to estimate this outcome measure. Outcome Definition 2 (adverse events) will define as follows: For the adverse event entry form, if all of the following conditions are met, it is defined as "liver disorder". (1) "Maralixibat (Livmarli)" has been selected as the drug to be administered. (2) "Yes" is selected for the presence or absence of adverse events due to the administered drug. (3) "Liver impairment and liver failure" are selected as symptoms/findings due to the administered drugs. (4) Date of occurrence or discovery of adverse event within the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/